CLINICAL TRIAL: NCT04504266
Title: Perioperative Optimization With Enhanced Recovery: The Effect of Health Habits on Surgical Outcomes in Patients Undergoing Major Abdominal Operations
Brief Title: Perioperative Optimization With Enhanced Recovery
Acronym: POWER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cindy Kin, Assistant Professor of Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 51827
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Complication of Surgical Procedure
Keywords: prehabilitation, exercise, nutrition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Recommendations to follow Mediterranean diet and exercise regularly before surgery.
- Prehab (Experimental): This intervention consists of a motivational interview and a mobile-app based coaching program to encourage patients to exercise and adopt a Mediterranean diet in the 3+ weeks prior to surgery.
  Interventions: Behavioral: POWER

INTERVENTIONS:
Behavioral: POWER — This intervention consists of a motivational interview and a mobile-app based coaching program to encourage patients to exercise and adopt a Mediterranean diet in the 3+ weeks prior to surgery.
  Arms: Prehab

SUMMARY:
This is a randomized controlled trial examining the effect of a motivational interview and perioperative mobile-app based nutrition and exercise intervention on surgical outcomes. The hypothesis is that such an intervention will improve surgical outcomes. Patients who are planned to undergo major elective abdominal surgery will be randomized to standard care or the nutrition/exercise intervention. This intervention consists of a mobile-app based coaching program to encourage patients to exercise and adopt a Mediterranean diet in the 3+ weeks prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* major abdominal surgery in 3+ weeks
* English or Spanish speaking

Exclusion Criteria:

* Unable to use smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical Complications occurring in the 90 day post-operative period, measured by the comprehensive complication index | 90 days after surgery
  The comprehensive complication index is an integrated score from 0 to 100 of all complications occurring in a specified time period and their severities as categorized by Clavien-Dindo classification. Calculation of the CCI is via a web-based calculator (www.assessurgery.com).

SECONDARY OUTCOMES:
Change in 6 minute walk test | It will take about 6 minutes to assess, and this will be performed at enrollment, right before surgery, and at 30 and 90 days after surgery
  Participants will be asked to walk as fast they can for 6 minutes using a validated mobile application (Timed Walk) to measure the distance walked.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Kin, MD, Principal Investigator — Stanford University; Brendan Visser, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kimura C, Liu Y, Crowder SE, Arbaugh C, Mai U, Shankar K, Shelton A, Visser B, Kin C. Barriers and Facilitators of Surgical Prehabilitation Adherence from the Patient Perspective: a Mixed Method Study. J Gastrointest Surg. 2023 Nov;27(11):2547-2556. doi: 10.1007/s11605-023-05857-9. Epub 2023 Oct 17. PMID 37848690